CLINICAL TRIAL: NCT07354087
Title: Impact of Molecular Pathological And Clinical Features for Adjuvant Treatment Selection in Endometrial Cancer: Multicentric Asian Registry (IMPACT-Endo-Asia)
Brief Title: Impact of Molecular Pathological And Clinical Features for Adjuvant Treatment Selection in Endometrial Cancer: Asian Registry
Acronym: IMPACTEndoAsia
Status: Active, not recruiting | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Supriya Sastri (chopra), Professor, Radiation Oncology, Tata Memorial Hospital
Other Study IDs: TMC IEC No 4453
Record Dates: First submitted 2025-01-24; First posted 2026-01-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The treatment practices for endometrial cancer have significantly changed over the last two decades. Nowadays, in addition to standard pathology, additional tests are performed to understand the behaviour of tumour so that personalized treatment can be advised for every patient. This approach ensures that patients with good cancer cell features receive minimum essential radiotherapy or surgery treatment with fewer side effects, while those with poor cell features undergo more aggressive treatment to improve their chances of survival.

However, this approach is not widely adopted in Asian countries. To address this, investigators are launching a project to gather data from various hospitals across Asia. The project aims to understand how different cancer cell factors impact treatment decisions and identify better ways to select additional treatment plans based on a patient's cancer cell features.

The project will gather data from around 250-300 patients who were evaluated or treated between January 2021 and December 2023. It will run for two years to improve our understanding and gain insights into the best ways to treat endometrial cancer.

DETAILED DESCRIPTION:
Endometrial cancer (EC) is the second most common gynecological malignancy affecting women worldwide. As per GLOBOCAN data, the incidence was 382,069 with a mortality of 89,929 in 2018, out of which Asia accounts for 40% of the new cases. By 2040 global incidence is predicted to increase by more than 50% as per the International Agency for Research on Cancer. Although the incidence is higher in the Western world, there is a persistent rising trend among low- and middle-income countries. EC is the fourth most common cause of cancer death among women of low socioeconomic status .3-5% of patients have inherited (Mismatch repair) mutation and are diagnosed to have Lynch syndrome also suggesting an overlapping genetic predisposition. Historically Bokhman's dualistic EC histopathological classification was based on tumor biological behavior and prognosis. Type I (60-70%) included endometrioid histology with a 5-year overall survival (OS) of 83-88%. The rest of the non-endometrioid histology was included in Type II (30%) which was associated with a higher risk of relapse and showed a 5-year OS of 54-64%. This classification had limited risk stratification, which led to inter-observer error of 60% and poor reproducibility of patient outcomes when references to pathological subtypes. Later two-tier tumor grading systems as per the International Federation of Gynecology and Obstetrics (FIGO) defined criteria had combined Grade 1 and 2 EC as low grade and Grade 3 EC as high grade. Several other high-risk features like myometrial invasion (MI) of more than 50%, substantial lymph vascular space invasion (LVSI), lymph node involvement, and tumor size of more than 2 cm were also considered in the classification. Prognostic classification based on morphological features alone leads to inaccuracies in tumor biology characterization, non-reproducibility due to the overlap of clinical-genetic characteristics causing heterogeneous molecular groups, heterogenous adjuvant treatment decisions (due to pathology variation).

More recently developments in genetics and molecular characterization have integrated classification methods, which include genomic profiling along with histopathological features. The Cancer Genome Atlas (TCGA)molecular classification first described four distinct subgroups based on molecular features which estimated the recurrence risk and predicted the survival in serous and endometrioid EC.

1. Pole ultra mutated (mutation in exonuclease domain of DNA polymerase epsilon)
2. Hypermutated with MSI/MMRd (loss of Mismatch Repair protein immunoreactivity)
3. Somatic copy number-low with frequent PI3K and WNT signaling abnormality (endometrioid-like)
4. Somatic copy number-high with frequent pathological variants in TP53(serous-like)

This molecular classification when integrated with standard pathology provided a relatively clearer distinction of outcomes.

Key observations from molecular classification studies also looking into clinical outcomes were as follows:

1. POLE mutation groups have shown consistently excellent outcomes and may benefit from the de-escalation of adjuvant therapy. However, no prospective results from randomized trials are yet available.
2. MMR/MSI status in metastatic EC can guide to select patients who can benefit from immunotherapy thus acts as a predictive biomarker for response to immunotherapy. The non-metastatic EC group has an intermediate prognosis but shows minimal benefit with adjuvant chemotherapy and radiotherapy. It is also used as a screening test for LS (hereditary nonpolyposis colorectal cancer).
3. Copy number low groups show a frequent mutation in the CTNNB1 gene. This group has over-expression of progesterone receptors (PR).
4. Copy number high (Serous EC and high-grade endometrioid EC) has frequent p53 mutations and poor outcomes are stage independent due to intrinsic aggressive biology. This group showed greater benefit with adjuvant chemotherapy. Improved outcomes have been observed when bevacizumab was added along with chemotherapy. This group also has low estrogen receptors (ER/PR) levels.

To simplify further and also to decrease the cost of diagnostic testing of molecular subgroups, the ProMisE study used surrogate markers to classify EC into four subgroups: POLEmut, MMR-d, p53wt and p53abn. The p53wt group does not harbor POLE/MMR-d/p53 mutation, so it is also termed as 'No Specific Molecular Profile (NSMP)'. The L1 neuronal Cell adhesion molecule(L1-CAM) is an independent prognostic marker as its upregulation is associated with the epithelial to mesenchymal transition (EMT), cell migration, cell invasion and thus its presence guides in patient selection for aggressive therapies due to their aggressive biology.

With the recent ESGO/ESTRO/ESP guideline update in 2021, there is a paradigm shift with integrated prognostic risk group stratification of EC patients which guides regarding the optimal management, that includes surgery, adjuvant therapy and surveillance recommendations. It also recommends treatment options when molecular classification is not available, as till today many centers have limited access to it. But there is a Heterogenous slow adaptation of molecular based classification in making adjuvant treatment decisions. Molecular profile-based classification has demonstrated prognostically valuable in Intermediate, High Intermediate and High-risk EC patients. The updated FIGO 2023 staging suggest for complete molecular classification in all endometrial cancers, which provide a better understanding of biological behaviors in EC.

While there are rapid transitions in recommendations based on Integrated molecular risk group stratification, most of the data on EC management originates from Europe and the USA. Asian region consists of different populations with different socio-economic statuses, variable access to medical infrastructure facilities, and availability of molecular profiling. This causes heterogeneous tissue reporting and impacts treatment decisions and future clinical trials.

The aim of registry is for better understanding the availability histopathological, Molecular subtyping and immunohistochemistry in Asian Institutes and its impact on adjuvant treatment decisions.

Patients evaluated or treated between January 2021 to December 2023 will be eligible for study participation and will be included in the study as per eligibility criteria.

Descriptive statistics (means, distributions) will be used for descriptive analysis. Log-rank test and cox-proportional hazard will be used for analysis of known prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

- Patients who were diagnosed to have EC and have access to standard histopathological reports and availability of treatment decisions.

Exclusion Criteria:

- Patients with final histopathological diagnosis of any other gynecological malignancy other than EC and its subtypes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We aim to include all patients with histological proven Endometrial Cancer from participating Institutes fulfilling the study criteria. This will allow better understanding of standard histopathological reporting and its impact on adjuvant treatment decisions.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-11-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
To study the Clinico-pathological characteristics in Endometrial Cancer | 24 months
  Proportion of Endometrial Cancer Molecular Subtypes (POLEmut, MMR-deficient, NSMP, p53 abnormal) and distribution of adjuvant radiation therapy types received (vaginal brachytherapy, external beam radiation therapy [EBRT], or combined radiation with chemotherapy) reported at treatment completion.
To study molecular characteristics in Endometrial Cancer. | 24 Months
  Proportion of Endometrial Cancer Cases by Tumor Grade, Histological Type, and Tumor Stage
To study the Clinicopathologic characteristics impact on treatment decision making across Asian regions | 24 Months
  proportion of patients who exhibit predefined clinicopathologic characteristics with percentages reported for each participating Asian region
To study molecular characteristics impact on treatment decision making across Asian regions. | 24 Months
  Proportion of participants whose treatment decisions are influenced by molecular characteristics. Data will be summarized by Asian region and analyzed in relation to clinical and demographic characteristics to assess the overall impact on treatment decision making.

SECONDARY OUTCOMES:
Comparison of risk grouping using standard histopathological features versus standard histopathological features plus molecular profile | 24 Months
  Percentage of patients grouped by risk using only standard pathology compared to risk groups based on both pathology and molecular test results, showing how often the groups match and how it affects predicting patient outcomes.
To report the selection of adjuvant treatment based on standard histopathological features alone or along with molecular risk features | 24 Months
  Percentage of participants who receive radiation and/or chemotherapy, categorized by documented risk-assessment method. Data will be collected via structured review of pathology, molecular test, and treatment records. Reported metric: proportion (%) in each risk-assessment group
To study the transition of staging towards FIGO 2023. | 24 Months
  Proportion of patient clinically stage using FIGO 2023 between 2 years.
To study the adequacy of risk grouping practices across Asian regions by comparing to ESTRO/ESGO/ESP and FIGO updates | 24 Months
  To study proportion of patient allocated across risk group using ESTRO VS FIGO 2023 guidelines.
To study the choice of External beam radiotherapy technique and brachytherapy applicators utilized | 24 Months
  Proportion of Patient receiving IMRT 3DCRT or Vaginal brachytherapy furthermore type of applicator used for brachytherapy.
To report the 3 years disease free survival | From the date of treatment completion till the date of any signs of recurrence / relapse upto a period of 3 years
  For Recruited participant disease free survival the time period between diagnosis to any relapse or last follow up or death due to any cause.
To study the family history in Endometrial Cancer | 24 Month
  Any history of a genetic curves in the family up to 3 generations of the family
To report the 3 years Local control. | From the date of treatment completion till the date of any signs of local control upto a period of 3 years
  Local control is time between diagnosis and local relapse and lost to follow up

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Sastri (Chopra), MD, DNB, Principal Investigator — ACTREC, Tata Memorial Centre
Locations (2):
- India (2):
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Advanced Centre for Treatment, Research and Education in Cancer, Tata Memorial Centre, Navi Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No